CLINICAL TRIAL: NCT07093229
Title: Gait Analysis as a Measure of Physical Performance in Managing Bilateral Knee Osteoarthritis in Elderly People
Brief Title: Knee Osteoarthritis in Elderly People - Gait Analysis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Diana Kamal (Other)
Responsible Party: Sponsor-Investigator, Diana Kamal, PhD, Filantropia Hospital
Organization: Filantropia Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Filantropia Hospital
Record Dates: First submitted 2025-07-14; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis; Physical Performance Parameters; Ultrasound; Quality of Life (QOL)
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Gait Analysis; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Experimental: Study Group. Elderly participants diagnosed with bilateral KOA will receive complete rehabilitation program (10 sessions of electrotherapy measures - transcutaneous nerve stimulation, ultrasound and low intensity laser treatment; 6 weeks of kinetic measures and gait training). Previous, all participants will be complete gait clinical, ultrasound and functional assess.
  Interventions: Other: Ultrasound exam of quadriceps muscles (left/right) and gait analysis; Other: Electrotherapy measures: transcutaneous nerve stimulation, ultrasound and low intensity laser; each one daily , applied on both lower limbs, for 10 days. Kinetic measures daily; Other: Gait training
- Control Group (Active Comparator): Active Comparator: Control Group Control Group will receive only 10 sessions of electrotherapy (transcutaneous nerve stimulation, ultrasound and low intensity laser treatment) and 6 weeks of kinetic measures, without gait control training. Previous, all participants will be complete clinical gait, ultrasound and functional assess.
  Interventions: Other: Ultrasound exam of quadriceps muscles (left/right) and gait analysis; Other: Electrotherapy measures: transcutaneous nerve stimulation, ultrasound and low intensity laser; each one daily , applied on both lower limbs, for 10 days. Kinetic measures daily

INTERVENTIONS:
Other: Ultrasound exam of quadriceps muscles (left/right) and gait analysis — Ultrasound exam (initial and after 3 months) - with SonoScape S9Pro; the investigators exam the thickness of the quadriceps muscle group between the superficial fat-muscle interface and the cortex of the femur and calculate the quadriceps muscle index as sum of both muscle thickness RT and LT cm/height2 (m2). The exam is conducted by a qualified sonographer. The examination is carried out on a one-on-one basis in a private setting where only the participant and the sonographer are present.
  Gait analysis with wireless system - BTS G-WALK; the investigators consider four gait parameters: Timed Up-and-Go (TUG) test, Symmetry index, Six Minutes Walking Test (6 MWT), and Walk cadence or average cadence (steps/min).
  Other Names: Electrotherapy measures; Kinetic program; Gait analysis; Functional assessment
Other: Electrotherapy measures: transcutaneous nerve stimulation, ultrasound and low intensity laser; each one daily , applied on both lower limbs, for 10 days. Kinetic measures daily — The gait training is the distinguish aspect in rehabilitation program. Usually, KOA training include only kinetic measures, without gait control training
  Other Names: Gait training
Other: Gait training — This type of special kinetic training includes Frenkel exercises for lower limb muscles and virtual / mirror exercises for different types of gait
  Arms: Study Group

SUMMARY:
The investigators perform a prospective controlled study and assess gait parameters in bilateral knee osteoarthritis (KOA) elderly patients with wireless system - BTS G-WALK, pre- and post-rehabilitation program. The complete assessment include: ultrasound exam, gait parameters and functional scale.

The investigators investigate the real impact of complete rehabilitation program, with gait control, on the physical performance and functional status.

ELIGIBILITY:
Inclusion Criteria:

* participants older than 65 years diagnosed with KOA according to ACR criteria, also accepted in our country;
* at least 5 years of disease progression;
* painful knee for a period of 48 hours after physical activity;
* absence of knee injuries at least 6 months before;
* absence of major disturbances in the frontal plane alignment of the knee;
* participants with other co-morbidities, but well controlled, like: arterial hypertension, dyslipidaemia and mellitus diabetes type II; a history of a symptomatic or complicated upper gastro-intestinal ulcer;
* compliance with physical exercise during the healthcare program.

Exclusion Criteria:

* unstable medical conditions preventing the patient from participating in the rehabilitation programs,
* history of knee replacement,
* neurological or any other conditions affecting strength or function of lower limbs.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Physical performance - gait analysis | 3 months
  Timed Up-and-Go (TUG) test (seconds) - participants stood up from an armed chair, walked at a safe and comfortable pace to a line 3 m away, crossed the line, turned, and returned to a sitting position in the chair; none of the patients used a walking aid and the time to complete the task was recorded.
Physical performance - gait analysis | 3 months
  Six Minutes Walking Test (6 MWT) - "walking distance" (meters) and "average cadence" (steps/minute).

SECONDARY OUTCOMES:
Functional status - quality of life | 3 months
  WOMAC scale contains 24 specific questions divided into three domains: pain (P-WOMAC; 5 items), stiffness (S-WOMAC; 2 items) and physical function (PF-WOMAC; 17 items). The score of each question ranges from 0 to 4. The 0 score is equivalent to maximal functional status and high scores 96 indicates a minimum status, with high disruption in day to day tasks.

OTHER OUTCOMES:
Quadriceps muscle index | 3 months
  In ultrasound exam, after establishing the midway point between the tip of the greater trochanter and the lateral joint line of the knee, the investigators identify the muscle tissue; the thickness of the quadriceps muscle (in centimeters) is established by measuring the space between the cortex of the femur and therefore the most superficial muscular fascia. Quadriceps muscle index is calculated as sum of both quadriceps muscle thickness Right and Left centimeters/ participant square height (square meters). Participant is exam with the knee extended.
Physical performance - gait analysis. Symmetry index | 3 months
  Symmetry index - for the participant's ability to have an identical model of acceleration and deceleration of their center of mass regardless of the side of the gait cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Diana Kamal, Craiova, Romania

IPD SHARING:
Plan to Share IPD: Undecided